CLINICAL TRIAL: NCT05005052
Title: Efficacy and Safety of Sulodexide in the Treatment of Chronic Primary Venous Disease of the Lower Extremities: A Randomized Placebo-Controlled Double-Blind Clinical Trial
Brief Title: Sulodexide in the Treatment of Chronic Primary Venous Disease of the Lower Extremities
Acronym: SuloPrima
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Value Outcomes Ltd. (Other)
Collaborators: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-002311-64
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Chronic Venous Disease; Chronic Insufficiency Venous
Keywords: sulodexide; venoactive drug; venous disease; randomized; blinded; CEAP; ultrasonography; angiology; conservative treatment; quality of life; productivity loss; EQ-5D; CIVIQ-20

STUDY DESIGN:
Intervention Model Description: two arms - the sulodexide arm compared to placebo arm
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulodexide arm (Experimental): Name: Vessel (medicinal product registered in Italy) Dosage form: soft capsules Active substance: sulodexidum 250 LSU Dosage: 2 x 2 soft capsules daily (oral use), in line with the labelled posology (500 LSU twice a day) Duration: 24 ± 4 weeks
  Interventions: Drug: Vessel
- Placebo arm (Placebo Comparator): Dosage form: soft capsules Appearance: undistinguishable from the active Dosage regimen: 2 x 2 soft capsules daily Duration of placebo intake: a total of 24 ± 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vessel — Sulodexide has protective effect on the endothelium, antithrombotic, fibrinolytic and anti-inflammatory effects. In the last 20 years, it has been well established in the common practice and its efficacy and safety have been demonstrated notably in the treatment of venous diseases such as post-thrombotic syndrome of the lower extremities, secondary prevention of deep and superficial venous thrombosis, supportive treatment of leg venous ulceration, ischemic disease of the lower limbs; symptomatic therapy of intermittent claudication, treatment of diabetic ulcers and microcirculation disorders of various aetiology. Patients with CVD were shown to respond quickly to sulodexide therapy in single arm observational studies. Sulodexide seems to provide both symptomatic and causal therapy.
  Arms: Sulodexide arm
Drug: Placebo — Placebo and no compression or venopharmaceutical regimen
  Arms: Placebo arm

SUMMARY:
This study compares the efficacy and safety of sulodexide (Vessel) to placebo in patients with chronic venous disease of the lower extremities.

The primary hypothesis is that more patients will achieve a decrease in rVCSS score of at least 4 points with sulodexide than with placebo.

DETAILED DESCRIPTION:
Chronic venous disease (CVD) prevalence is increasing in developed countries. The frequency reported in different sources ranges between 10 and 50% of the population and its rise is expected resulting from the overall aging of the population. The most common symptoms of Chronic venous disease of lower extremities include, increased limb fatigue, heaviness and swelling, pain, cramps, itching, and trophic skin changes that can result in a venous ulcer. CVD has a significant impact on the patient's quality of life and their work productivity.

Conservative treatment consists of lifestyle measures, compression therapy and use of venoactive drugs (venopharmaceuticals). Venoactive drugs are a heterogenous group of compounds with various mechanisms of action, such as increasing venous wall tonus, reducing capillary fragility and permeability, increasing capillary resistance, and improving lymphatic drainage. The goal of the treatment is anti-oedematous action, improvement of trophism of affected tissues, reduction of subjective symptoms, swelling of the limbs and affecting related trophic skin changes which leads to the increase of quality of life.

Sulodexide has protective effect on the endothelium, antithrombotic, fibrinolytic and anti-inflammatory effects. In the last 20 years, it has been well established in the common practice and its efficacy and safety have been demonstrated notably in the treatment of venous diseases such as post-thrombotic syndrome of the lower extremities, secondary prevention of deep and superficial venous thrombosis, supportive treatment of leg venous ulceration, ischemic disease of the lower limbs; symptomatic therapy of intermittent claudication, treatment of diabetic ulcers and microcirculation disorders of various aetiology. Patients with CVD were shown to respond quickly to sulodexide therapy in single arm observational studies. Sulodexide seems to provide both symptomatic and causal therapy. The aim of the present study is to provide the first high-level (causal) evidence on the efficacy and safety of sulodexide across the whole spectrum of patients suffering from symptomatic primary CVD (CEAP classification C2S to C6S).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed primary venous disease of the lower limbs in stage C2 - C6 according to the CEAP classification, clinical involvement of the venous system of the lower limbs is verified by duplex ultrasonography
* Presence of objective and subjective symptoms of the disease (classified according to rVCSS score ≥ 4)
* At the time of the enrolment, patient is not using nor planning to use compression therapy from his own decision or the decision of the treating physician
* The patient signed an informed consent for inclusion in the clinical trial and consent to the processing of personal data
* Patient over 18 years of age
* Male or female patient of non-childbearing potential, i.e.: post-menopausal (at least 2 years without spontaneous menses) or surgically sterile (bilateral tubal occlusion or hysterectomy or ablation of both ovaries); OR of childbearing potential but with a negative pregnancy test result at Visit 1 AND agrees to use a highly effective method of contraception

Exclusion Criteria:

* Use of a drug with venoactive effect in the last month
* Regular use of compression therapy or use of mechanical devices for reduction of oedema in the last month
* Heart Failure as per NYHA III and IV, congestive heart failure with peripheral oedemas
* Chronic kidney disease with GF < 30 ml/min (< 0,5 ml/s) and/or proteinuria > 0,5 g/24 hours, nephrotic syndrome, renal oedemas
* Advanced liver disease (Child-Pugh B and C or laboratory values of ALT or AST more than 3 times upper limit of normal range)
* Deep venous thrombosis lower limb thrombosis and / or documented residual venous obstruction or deep venous reflux due to post-thrombotic changes in the deep venous system
* Superficial venous thrombosis of the lower limbs in the previous 6 months
* Congenital venous / venolymphatic venous malformation
* Neuropathy of any aetiology
* Diabetic foot syndrome
* Refractory (uncontrollable) arterial hypertension (inability to achieve therapeutically systolic blood pressure ≤ 160 mmHg or diastolic blood pressure ≤ 100 mmHg)
* Symptomatic ischemic disease of lower limbs
* Lymphoedema: primary, posttraumatic, postoperative, post-radiation, malignant
* Manual/instrumental lymphatic drainage in the last 6 months
* Invasive procedure on the lower limbs in the last 6 months
* Trauma of the lower extremity that has not fully healed
* Use of oral/parenteral anticoagulants, dual antiplatelet therapy, diuretics, corticosteroids, oestrogens, or progesterone and its derivates
* Chronic pain treatment ≥ 14 days
* Psychopharmaceuticals affecting fluid retention (antipsychotics, combined antidepressants)
* Pathologic obesity (BMI > 40 kg/m2)
* The patient is currently enrolled in another interventional or non-interventional study
* Contraindications to the administration of sulodexide according to IB (haemorrhagic diathesis, hypersensitivity to the drug substance or any of the excipients, heparin, heparinoids or other glycosaminoglycans (GAGs), etc.)
* Patients with active malignant disease or malignant disease in remission for less than 5 years
* Pregnancy
* Breastfeeding

Continuous exclusion criteria:

* Clinically significant progression of the investigated condition, which requires urgent or early invasive therapy (as assessed by the investigating physician)
* Onset of any condition requiring initiation of the not permitted medication/treatment
* Serious adverse reactions
* Pregnancy

Compression therapy can be initiated anytime during the trial participation in case that patient experiences worsening of the rVCSS score of at least 4 points compared to baseline AND the treating physician decides to prescribe such regimen. Certified/notified compression stockings of class II (23-32 mmHg) based on circular knit are allowed. Patients initiating compression therapy are not excluded but the stocking need to be taken off a day before the scheduled study visit. The treatment allocation in patients initiating compression therapy remain blinded.

In case compression therapy is initiated during study participation, information about the date of initiation, type and adherence is collected in the following visits.

If sufficient proportion of subjects is switched to compression therapy, compression therapy will be tested as effect modifier across CEAP classes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Revised Venous Clinical Severity Score (rVCSS) | 24 weeks of treatment
  A minimal decrease in rVCSS score by 4 points will be considered a clinically significant response to treatment.

SECONDARY OUTCOMES:
Revised Venous Clinical Severity Score (rVCSS) | 4, 8 and 12 weeks of treatment
  A minimal decrease in rVCSS score by 4 points will be considered a clinically significant response to treatment.
Volume in lower limb | 4, 8, 12 and 24 weeks of treatment
  The decrease of lower limb volume of at least 30 mL will be determined using water displacement leg volumetry and will be considered a clinically significant response to treatment.
Visual Analogue Scale (VAS) | 4, 8, 12 and 24 weeks of treatment
  Decrease in mean pain on Visual Analogue Scale.
Work Productivity and Activity Impairment (WPAI questionnaire) | 8 and 24 weeks of treatment
  Increase in mean work productivity in WPAI questionnaire.
EQ-5D questionnaire | 8 and 24 weeks of treatment
  Increase in the mean generic quality of life in EQ-5D questionnaire.
Chronic Venous Insufficiency Quality of Life (CIVIQ-20 questionnaire) | 8 and 24 weeks of treatment
  Increase in the mean disease-specific quality of life in CIVIQ-20 questionnaire.
Mean time of clinically significant worsening rVCSS | 4, 8, 12 and 24 weeks of treatment
  Mean time of worsening the rVCSS score since study initiation of at least 4 points. The difference will be visualized using Kaplan-Meier estimates and tested using Cox proportional-hazards models.
Compression therapy initiation | 4, 8, 12 and 24 weeks of treatment
  Mean time of duration of initiation of compression therapy since study initiation. The difference will be visualized using Kaplan-Meier estimates and tested using Cox proportional-hazards models.

CONTACTS AND LOCATIONS:
Locations (19):
- Czechia (19):
  - CardioVasc s.r.o., Mladá Boleslav, Central Bohemia
  - Oblastní nemocnice Mladá Boleslav, a.s., Mladá Boleslav, Central Bohemia
  - Phlebomedica s.r.o., Říčany, Central Bohemia
  - Angionika s.r.o., Slaný, Central Bohemia
  - Cor et Vasa s.r.o, Český Těšín, Moravskoslezský kraj
  - Angiologická ambulance s.r.o., Hlučín, Moravskoslezský kraj
  - Angiologie Opava s.r.o., Opava, Moravskoslezský kraj
  - Pedicor s.r.o., Ostrava, Moravskoslezský kraj
  - Péče o cévy s.r.o., Ostrava, Moravskoslezský kraj
  - Chirurgická ambulance MUDr. Prokop, Ostrava, Moravskoslezský kraj
  - Cordesora s.r.o., Olomouc, Olomoucký kraj
  - Angios s.r.o., Prostějov, Olomoucký kraj
  - REAGINTA sro, Přerov, Olomoucký kraj
  - CTC Hodonín s.r.o., Hodonín, South Moravian
  - MUDr. Jan KVASNIČKA,CSc., Ordinace pro choroby srdce a cév, Prague
  - Žilní klinika, Prague
  - FLEBODERMA, s.r.o., Prague
  - Cévní ambulance - Poliklinika Modřany, Prague
  - MUDr.Simon Jirát s.r.o. - Angiologie Zbraslav, Prague

IPD SHARING:
Plan to Share IPD: Undecided